CLINICAL TRIAL: NCT03390621
Title: Parental Feeding Styles and Child Dietary Quality at Dinner Among Low-income Minority Families
Brief Title: Parental Feeding Styles and Child Dietary Quality
Status: Completed | Type: Observational
Sponsor: Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Sheryl Hughes, Associate Professor, Baylor College of Medicine
Other Study IDs: 18541HEI
Record Dates: First submitted 2017-12-21; First posted 2018-01-04 (Actual); Last update posted 2018-01-04 (Actual); Status verified 2017-12

CONDITIONS: Dietary Quality
Keywords: parent feeding styles; dietary quality; dinner meal; preschool; low-income

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In this study, the investigators will use an existing data set to examine the relationship between parent feeding styles and the quality of the dinner meal using the Healthy Eating Index.

DETAILED DESCRIPTION:
Investigators will use an existing data set collected between 2007 and 2009. The purpose of the larger data set including 177 families was to examine parent - child interactions during dinner meals in low-income Hispanic and African-American families participating in Head Start programs. Data was collected on parent-child interactions and information regarding the food served and consumed by children during dinner meals. The specific aims included: 1) examining the overall diet quality using the Healthy Eating Index of Head Start preschool dinner meals by parent feeding styles, an 2) the diet quality of the dinner meal served to that of the meal consumed and within each of the parent feeding styles.

ELIGIBILITY:
Inclusion Criteria:

* Parents who were responsible for feeding the child while the child was not in Head Start and their oldest child enrolled in Head Start.

Exclusion Criteria:

* Any children who have dietary restraints or food allergies.

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Individuals from the larger data set of 177 families who had complete dietary and demographic data.
Sampling Method: Non-Probability Sample
Enrollment: 177 (Actual)
Dates: Start 2007-01-01 (Actual); Primary Completion 2009-02-28 (Actual); Study Completion 2009-12-31 (Actual)

PRIMARY OUTCOMES:
Dietary Quality | 10 minutes
  The Healthy Eating Index was used to obtain the quality of the food served and consumed by the child at dinner.

CONTACTS AND LOCATIONS:
Overall Officials: Sheryl O Hughes, PhD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hughes SO, Power TG, Papaioannou MA, Cross MB, Nicklas TA, Hall SK, Shewchuk RM. Emotional climate, feeding practices, and feeding styles: an observational analysis of the dinner meal in Head Start families. Int J Behav Nutr Phys Act. 2011 Jun 10;8:60. doi: 10.1186/1479-5868-8-60. PMID 21663653